CLINICAL TRIAL: NCT02714998
Title: The Impact of Salpingectomy and Single Dose Systemic Methotrexate Treatments on Ovarian Reserve in Ectopic Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Enes Taylan, Medical Doctor, Ob&Gyn Specialist, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-TIP-043
Record Dates: First submitted 2016-03-14; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Ectopic Pregnancy; Infertility
Keywords: ectopic pregnancy; ovarian reserve; salpingectomy; methotrexate
MeSH Terms: conditions — Pregnancy, Ectopic; Infertility | interventions — Methotrexate; Salpingectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methotrexate only (Active Comparator): Single dose of systemic Methotrexate administered to 55 patients.
  Interventions: Drug: Methotrexate
- Salpingectomy only group (Active Comparator): Laparoscopic unilateral salpingectomy performed to 61 patients.
  Interventions: Procedure: salpingectomy
- Salpingectomy following Methotrexate (Active Comparator): 15 patients underwent laparoscopic unilateral salpingectomy following unsuccessful single dose of methotrexate administration.
  Interventions: Drug: Methotrexate; Procedure: salpingectomy

INTERVENTIONS:
Drug: Methotrexate — single dose systemic methotrexate administration (50 mg/m2)
  Other Names: Mtx
  Arms: Methotrexate only; Salpingectomy following Methotrexate
Procedure: salpingectomy — Laparoscopic unilateral salpingectomy
  Arms: Salpingectomy following Methotrexate; Salpingectomy only group

SUMMARY:
The investigators aimed to investigate the effects of salpingectomy and Methotrexate administration on ovarian reserve in ectopic pregnancy.

DETAILED DESCRIPTION:
In this study, the effects of unilateral laparoscopic salpingectomy and single dose of systemic Methotrexate administration on ovarian reserve in patients diagnosed with ectopic pregnancy were investigated.

ELIGIBILITY:
Inclusion Criteria:

* ectopic pregnancy diagnosis

Exclusion Criteria:

* history of endometriosis, ovarian surgery, systemic chemotherapy, ART treatment.
* patients treated with multiple doses of methotrexate or different surgical procedure (salpingostomy, milking)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve assessment by measuring AMH level. | 1-3 months
  Ovarian reserve were assessed before and after treatment by measuring AMH levels.

SECONDARY OUTCOMES:
Number of participants with treatment related adverse effect on fertility. | 2 years of follow up after treatment
  Rates of term delivery, spontaneous abortion, recurrent ectopic pregnancy and ongoing pregnancy for each group of patients were calculated during 2 years of follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet M. Ergenoglu, Ass. Prof., Study Director — Ege University School of Medicine Department of Obstetrics and Gynecology
Locations (1):
- Ege University School of Medicine Department of Obstetrics and Gynecology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to share patient data yet. However, it is possible if approved by ethical committee.